CLINICAL TRIAL: NCT03375125
Title: Safety and Efficacy of L. Reuteri ATCC PTA 5289 & L. Reuteri DSM 17938 in Pregnant Women to Improve Oral Health and Reduce the Risk for Prematurity or Intrauterine Growth Retardation (IUGR)
Brief Title: L. Reuteri ATCC PTA 5289 + L. Reuteri DSM 17938 in Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: University of Bari (Other); BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Research on Translational Research Center on Mother-Child Health, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0138
Record Dates: First submitted 2017-11-29; First posted 2017-12-15 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis and Pregnancy
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind allocation concealment, parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization list will by assembled by independient organization not related with participant, care provider, investigators or sponsors. eCRF will include randomization selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): L. reuteri DSM 17938 + L. reuteri ATCC PTA 5289), dose of 2x10^8 Colony Forming Units (CFU). One lozenges will be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo will have identical appearance, taste, and flavor, except for lacking the bacteria. One lozenges will be taken twice per day (one in the morning and one in the afternoon)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — L. reuteri DSM 17938 & L. reuteri ATCC PTA 5289 ) will be given at a dose of 2x10^8 Colony Forming Units (CFU). One lozenges is to be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day.
  Arms: Probiotic
Other: Placebo — Placebo will have identical appearance, taste, and flavor, except for lacking the bacteria. One lozenges will be taken twice per day (one in the morning and one in the afternoon)
  Arms: Placebo

SUMMARY:
Randomized controlled tril to evaluate the safety and efficacy for the combination of L. reuteri ATCC PTA 5289 & L. reuteri DSM 17938 in pregnant women with periodontitis and/or gingivits to improve oral health and at the same time reduce the risk for prematurity or intrauterine growth retardation (IUGR).

Women in this study wil receive L. reuteri Prodentis (L. reuteri DSM 17938 & L. reuteri ATCC PTA 5289 ) at a dose of 2x10^8 Colony Forming Units (CFU). One lozenges is to be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day since randomization until delivery. The control group will receive placebo lozenges which contains identical ingredients except for lacking the bacteria. One lozenges is to be taken twice per day (one in the morning and one in the afternoon. The study product will be kept refrigerated (+20 - +80 C)

DETAILED DESCRIPTION:
Rationale. Gingivitis and periodontitis represent highly prevalent oral pathologies in pregnant women. The physiological, immunological and endocrine changes imposed by pregnancy are associated with a greater predisposition for the development of gingivitis. Considering the potential association between the presence of gingivitis and the development of complications during pregnancy and the time of delivery (preeclampsia, preterm, IUGRs), it is important to evaluate the impact of early administration of a mixture of lactobacillus on improved health oral status, and at the same time assessing the effect on risk reduction of prematurity and/or IUGRs.

For primary outcome the investigators will evaluate the changes along the study in the oral health status evaluated through a composite of Modified Gingival Index (Lobene) + Plaque Index (Silnes and Loe) + Gingival Bleeding Index + Probing pocket depth (PPD) and Clinical attachment level (CAL).

For secondary outcomes the investigators will evaluate rate of prematurity and or Intrauterine growth retardation; changes in mother salivary markers of systemic inflammation; profile of inflammosome in placenta and new born cord blood; lactobacilli, bifidobacteria and streptococcus profile in vagina by RT-PCR (specific primers); changes during the study for oral microbiome Intervention group wil receive L. reuteri Prodentis (L. reuteri DSM 17938 & L. reuteri ATCC PTA 5289 ) at a dose of 2x10^8 Colony Forming Units (CFU). One lozenges is to be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day since randomization until delivery.

The control group will receive placebo lozenges which contains identical ingredients except for lacking the bacteria. One lozenges is to be taken twice per day (one in the morning and one in the afternoon. The study product will be kept refrigerated (+20 - +80 C)

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Age (Italy: 18-40 years; Mexico: 15-40 years)
* Gestational week (Mexico: >8 weeks and 16 weeks; Italy: >8 weeks and 12 weeks)
* Mild to Severe Gingival and Periodontal disease verified by dentist using Lobene Modified Gingival Index, Plaque Index, Gingival Bleeding Index, probing pocket depth (PPD) and clinical attachment level (CAL)
* Signed Informed consent

Exclusion Criteria:

* Pathologic pregnancy (except for preeclampsia and/or bacteriuria)
* Severe obesity (Body Mass Index>35)
* Use of any product containing probiotics 2 weeks before randomization
* Use of any product containing chlorhexidine 2 weeks before randomization
* Antibiotic therapy within 2 weeks before randomization
* Known allergies towards the ingredients of the experimental product
* Inability to comprehend to the study protocol
* Systemic diseases differnt that periodontal disease

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of periodontal disease | 6 months
  Changes along the study in periodontal disease evaluated through Modified Gingival Index

SECONDARY OUTCOMES:
Prematurity risk reduction | At delivery
  Rate of prematurity at moment of delivery
Mother Inflammosome profile | 6 months
  Changes in salivary biomarkers of inflammation
Placental Inflammosome | At delivery
  Profile of cytokines measured in placenta at delivery
Changes in vaginal microbiome | 6 months
  Measurement of vaginal lactobacilli, bifidobacteria and streptococcus microbiome by RT-PCR
Intrauterine growth retardation (IUGR) risj reduction | At delivery
  Rate of Intrauterine growth retardation (IUGR) at delivery
Newborn cord blood inflammosome | At delivery
  Profile of cytokines measured in new-born cord blood at delivery

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Pediatric. Università di Bari; Ospedale Pediatrico Giovanni XXIII, Bari, Italy
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krasse P, Carlsson B, Dahl C, Paulsson A, Nilsson A, Sinkiewicz G. Decreased gum bleeding and reduced gingivitis by the probiotic Lactobacillus reuteri. Swed Dent J. 2006;30(2):55-60. PMID 16878680
- [Result] Staab B, Eick S, Knofler G, Jentsch H. The influence of a probiotic milk drink on the development of gingivitis: a pilot study. J Clin Periodontol. 2009 Oct;36(10):850-6. doi: 10.1111/j.1600-051X.2009.01459.x. Epub 2009 Aug 12. PMID 19682173
- [Result] Harini PM, Anegundi RT. Efficacy of a probiotic and chlorhexidine mouth rinses: a short-term clinical study. J Indian Soc Pedod Prev Dent. 2010 Jul-Sep;28(3):179-82. doi: 10.4103/0970-4388.73799. PMID 21157050
- [Result] Slawik S, Staufenbiel I, Schilke R, Nicksch S, Weinspach K, Stiesch M, Eberhard J. Probiotics affect the clinical inflammatory parameters of experimental gingivitis in humans. Eur J Clin Nutr. 2011 Jul;65(7):857-63. doi: 10.1038/ejcn.2011.45. Epub 2011 Mar 30. PMID 21448219
- [Result] Iniesta M, Herrera D, Montero E, Zurbriggen M, Matos AR, Marin MJ, Sanchez-Beltran MC, Llama-Palacio A, Sanz M. Probiotic effects of orally administered Lactobacillus reuteri-containing tablets on the subgingival and salivary microbiota in patients with gingivitis. A randomized clinical trial. J Clin Periodontol. 2012 Aug;39(8):736-44. doi: 10.1111/j.1600-051X.2012.01914.x. Epub 2012 Jun 13. PMID 22694350
- [Result] Stensson M, Koch G, Coric S, Abrahamsson TR, Jenmalm MC, Birkhed D, Wendt LK. Oral administration of Lactobacillus reuteri during the first year of life reduces caries prevalence in the primary dentition at 9 years of age. Caries Res. 2014;48(2):111-7. doi: 10.1159/000354412. Epub 2013 Nov 29. PMID 24296746
- [Result] Toiviainen A, Jalasvuori H, Lahti E, Gursoy U, Salminen S, Fontana M, Flannagan S, Eckert G, Kokaras A, Paster B, Soderling E. Impact of orally administered lozenges with Lactobacillus rhamnosus GG and Bifidobacterium animalis subsp. lactis BB-12 on the number of salivary mutans streptococci, amount of plaque, gingival inflammation and the oral microbiome in healthy adults. Clin Oral Investig. 2015 Jan;19(1):77-83. doi: 10.1007/s00784-014-1221-6. Epub 2014 Mar 18. PMID 24638207